CLINICAL TRIAL: NCT07025876
Title: Evaluation of the Safety and Tolerability of 24-valent Pneumococcal Polysaccharide Conjugate Vaccine in Individuals Aged 18 Years and Above: A Random PhaseⅠClinical Trial
Brief Title: PhaseⅠClinical Trial of 24-valent Pneumococcal Polysaccharide Conjugate Vaccine
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Jiangsu Province Centers for Disease Control and Prevention (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: JSVCT182
Record Dates: First submitted 2025-06-06; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Streptococcus Pneumoniae Pneumonia
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Low-dose group (Experimental): Adults receive one dose of 0.5ml low-dose PCV24 vaccine.
  Interventions: Biological: low dose PCV24
- High-dose group. (Experimental): Adults receive one dose of 0.5ml high-dose PCV24 vaccine.
  Interventions: Biological: high dose PCV24
- Positive control group (Active Comparator): Adults receive one dose of 0.5ml PPV23 vaccine.
  Interventions: Biological: PPV23
- placebo control group (Placebo Comparator): Adults receive one dose of 0.5ml normal saline.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: low dose PCV24 — The 24-valent pneumococcal polysaccharide conjugate vaccine (low-dose) developed by Shanghai Ruizhou Biotechnology Co., Ltd. and Changchun Ruizhou Biopharmaceutical Co., Ltd. is a liquid formulation. Each vial contains 0.5 ml, with a dosage of 0.5 ml per person per administration. The polysaccharide content of each serotype is as follows:
  * 3 serotypes (3, 6B, 12F): 4.0 μg per vial each
  * 21 other serotypes (1, 2, 4, 5, 6A, 7F, 8, 9N, 9V, 10A, 11A, 14, 15B, 17F, 18C, 19A, 19F, 20, 22F, 23F, 33F): 2.0 μg per vial each After conjugation with carrier proteins, the polysaccharides of each serotype are adsorbed onto an aluminum phosphate adjuvant (aluminum content: 0.25 mg per dose).
  Arms: Low-dose group
Biological: high dose PCV24 — The 24-valent pneumococcal polysaccharide conjugate vaccine (high-dose) developed by Shanghai Ruizhou Biotechnology Co., Ltd. and Changchun Ruizhou Biopharmaceutical Co., Ltd. is a liquid formulation. Each vial contains 0.5 ml, with a dosage of 0.5 ml per person per administration. The polysaccharide content of each serotype is as follows:
  3 serotypes (3, 6B, 12F): 8.0 μg per vial each 21 other serotypes (1, 2, 4, 5, 6A, 7F, 8, 9N, 9V, 10A, 11A, 14, 15B, 17F, 18C, 19A, 19F, 20, 22F, 23F, 33F): 4.0 μg per vial each After conjugation with carrier proteins, the polysaccharides of each serotype are adsorbed onto an aluminum phosphate adjuvant (aluminum content: 0.25 mg per dose).
  Arms: High-dose group.
Biological: PPV23 — The 23-valent pneumococcal polysaccharide vaccine (PPV23) produced by Chengdu Institute of Biological Products is available in vials of 0.5 ml, with a dosage of 0.5 ml per person per administration. It contains the following pneumococcal polysaccharides for each serotype:
  Serotypes 1, 2, 3, 4, 5, 6B, 7F, 8, 9N, 9V, 10A, 11A, 12F, 14, 15B, 17F, 18C, 19A, 19F, 20, 22F, 23F, and 33F: 25 μg per vial for each serotype.
  Additionally, it contains sodium chloride and water for injection.
  Arms: Positive control group
Biological: Placebo — In addition to the antigen components, the 24-valent pneumococcal polysaccharide conjugate vaccine developed by Shanghai Ruizhou Biotechnology Co., Ltd. and Changchun Ruizhou Biopharmaceutical Co., Ltd. contains the following excipients:
  Aluminum phosphate adjuvant (aluminum content: 0.25 mg per dose) Sodium chloride Succinic acid Polysorbate 80 Water for injection It is a liquid formulation, available in vials of 0.5 ml, with a dosage of 0.5 ml per person per administration.
  Arms: placebo control group

SUMMARY:
In the treatment of pneumococcal diseases, the common use of penicillin-based antimicrobial agents has led to drug resistance, which has become a global challenge. Therefore, disease prevention through vaccination is essential. The 23-valent pneumococcal polysaccharide vaccine, the first widely used vaccine, has limitations. Subsequent pneumococcal polysaccharide conjugate vaccines have improved protection rates but increased cases of infections caused by non-vaccine serotype strains. Currently, vaccines available in China for pneumococcal disease prevention include the 23-valent polysaccharide vaccine (approved only for adults) and the 13-valent conjugate vaccine. PCV24 expands serotype coverage and converts capsular polysaccharides into T-cell-dependent antigens by binding them to proteins, stimulating humoral immunity and the complement system to generate specific antibodies and immunological memory for disease prevention. This study aims to preliminarily investigate the safety and immunogenicity of PCV24 vaccination in Chinese adults.

DETAILED DESCRIPTION:
Streptococcus pneumoniae is a Gram-positive diplococcus, and its capsular polysaccharide is a key virulence factor. According to differences in the composition and structure of capsular polysaccharides, it can be divided into more than 90 serotypes, with varying viability and pathogenicity among different serotypes. As an important opportunistic pathogen, this bacterium can breach mucosal defense systems to cause invasive infections when host immunity declines, leading to diseases such as pneumonia, bacterial meningitis, bacteremia, sinusitis, and otitis media.

Antimicrobial agents commonly used in the treatment of pneumococcal diseases, such as penicillins, macrolides, and cephalosporins, have faced global challenges due to drug resistance, making vaccination essential for disease prevention. The World Health Organization (WHO) has classified pneumococcal diseases as a top priority for vaccination. The early widely used 23-valent pneumococcal polysaccharide vaccine had limitations, while subsequent 7-valent, 10-valent, and 13-valent pneumococcal polysaccharide conjugate vaccines improved protection rates but were associated with increased infections from non-vaccine serotype strains. Currently, only the 23-valent polysaccharide vaccine is approved for adult use in China. Pneumococcal conjugate vaccines convert capsular polysaccharides into T-cell-dependent antigens by binding them to proteins, thereby stimulating humoral immunity and the complement system to generate specific antibodies and immunological memory for disease prevention. This study aims to evaluate the safety and tolerability of a 24-valent pneumococcal polysaccharide conjugate vaccine in individuals aged 18 years and older.

ELIGIBILITY:
Inclusion Criteria:

* 1.Age and Identification: Volunteers aged ≥18 years on the screening day, able to provide valid legal identification.

  2.Informed Consent: Volunteers who have received and understood the study information, voluntarily agreed to participate, and signed the Informed Consent Form.

  3.Compliance: Volunteers able and willing to adhere to the clinical trial protocol requirements and attend all scheduled visits.

  4.Baseline Temperature: Axillary temperature ≤37.0°C on the enrollment day.

Exclusion Criteria:

* 5.Vaccination History: Prior receipt of pneumococcal conjugate vaccine; pneumococcal polysaccharide vaccine within the past 3 years; or a history of invasive Streptococcus pneumoniae disease.

  6.Severe Allergic Reactions: History of severe allergic reactions, such as anaphylactic shock, allergic laryngeal edema, allergic purpura, thrombocytopenic purpura, local allergic necrotic reaction (Arthus reaction), etc.

  7.Immunocompromised Status: Diagnosed congenital or acquired immunodeficiency; or receipt of systemic glucocorticoid therapy (e.g., prednisone or equivalent >5 mg/day for ≥2 consecutive weeks) within 1 month prior to vaccination (local, inhaled, or nebulized steroids are permitted).

  8.Severe Cardiovascular Diseases: History of arrhythmia, conduction block, myocardial infarction, or uncontrolled severe hypertension (on-site measurement: systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥100 mmHg).

  9.Acute Illness or Medication Use: Acute febrile illness, acute infectious disease, active cold symptoms, progressive influenza, or current use of related therapeutic medications.

  10.Neurological/Developmental Disorders: History of neurological impairment, severe congenital malformation, severe developmental disorder, severe genetic defect, or severe malnutrition.

  11.Neuropsychiatric History: Personal or family history of epilepsy, encephalopathy, or psychiatric disorders.

  12.Coagulation Abnormalities: Diagnosed thrombocytopenia, coagulation dysfunction (e.g., coagulation factor deficiency, coagulation disorders, platelet abnormalities), or contraindications to intramuscular injection (e.g., anticoagulant therapy).

  13.Splenic Abnormalities: Asplenia, functional asplenia, or splenectomy for any reason.

  14.Uncontrolled Chronic Diseases: Severe chronic diseases or progressive conditions that cannot be stably controlled.

  15.Blood Products/Immunoglobulins: Receipt of blood or blood products, or immunoglobulins within the past 3 months.

  16.Live Attenuated Vaccines: Vaccination with live attenuated vaccines within the past 14 days.

  17.Other Vaccines: Vaccination with other vaccines within the past 7 days. 18.Investigational Products: Receipt of other investigational drugs or vaccines within the past 1 month.

  19.Concurrent Studies: Current participation or planned participation in another clinical study of drugs or vaccines during the research period.

  20.Investigator's Discretion: Any other condition that, in the investigator's judgment, may interfere with study evaluation.

  21.Additional Exclusions for Specific Populations: Females of Childbearing Potential (18-49 years): Positive urine pregnancy test on enrollment day; lactation; or planning to become pregnant within 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2023-11-18 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
To evaluate The incidence of adverse reactions after vaccination | Within 0-7 days after vaccination
  The proportion of subjects reporting adverse reactions within 7 days after vaccination

SECONDARY OUTCOMES:
To evaluate The incidenceof adverse events after vaccination. | Within 0-30 days after vaccination
  The proportion of subjects reporting adverse events within 0-30 days after vaccination.
To evaluate The occurrence of serious adverse events after vaccination. | Within 6 months after vaccination
  The proportion of subjects reporting serious adverse events after vaccination.
Number of participants with clinically significant changes in blood routine after vaccination | Day 3 after vaccination
  Changes in blood routine indicators on day 3 after vaccination
Number of participants with clinically significant changes in blood biochemistry after vaccination | Day 3 after vaccination
  Measurement: Changes in blood biochemistry indicators on day 3 after vaccination
Number of participants with clinically significant changes in coagulation function after vaccination | Day 3 after vaccination
  Changes in coagulation function indicators on day 3 after vaccination
Number of participants with clinically significant changes in urinalysis after vaccination | Day 3 after vaccination
  Changes in urinalysis indicators on day 3 after vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Provincial Center for Diseases Control and Prevention, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No